CLINICAL TRIAL: NCT02655744
Title: Prospective Neurobehavioral Outcomes Follow-up in Primary CNS Lymphoma Patients Treated With Cranial Radiotherapy Combined With or Without MTX-based Chemotherapy According to the Multidisciplinary Treatment Guidelines Implemented at a Single Institute
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-5392B
Record Dates: First submitted 2015-12-09; First posted 2016-01-14 (Estimated); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Primary Central Nervous System Lymphoma
Keywords: Neurobehavioral Assessment; Radiotherapy (RT); Chemotherapy; Neurotoxicity
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- newly-diagnosed patients with primary CNS lymphoma
  Interventions: Radiation: Standard treatment protocol with combined chemoradiation

INTERVENTIONS:
Radiation: Standard treatment protocol with combined chemoradiation

SUMMARY:
Background. Primary central nervous system lymphoma (PCNSL) is an uncommon disease. Conventional treatment has consisted of either whole brain radiotherapy (WBRT) or methotrexate (MTX)-based combined modality therapy combining chemotherapy and cranial irradiation. The treatment principles at our institute have been quite consistent in the past, sticking to the treatment protocol reported by Memorial Sloan-Kettering Cancer Center in 1990s. No matter what the dosage of MTX is, it is well-established that the addition of chemotherapy to cranial RT significantly improved survival outcomes. However, it was found that delayed treatment-related cognitive sequelae emerged as a significant debilitating complication of combined modality treatment in patients with PCNSL, especially when effective treatment can achieve disease control and better survival rates. Furthermore, the specific contribution of the disease per se and various treatment modalities to cognitive impairment remains to be clarified because the neurotoxic potential of combined modality treatments is difficult to differentiate when each can result in cognitive dysfunctions respectively.

Treatment-related neurotoxicity could be demonstrated by virtue of several meaningful indicators, including neurobehavioral assessments, neuroimaging outcomes, and even measures of quality-of-life (QoL).

Methods. Therefore, this one-year individual research will be a prospective observational cohort study with a longitudinal assessment of neurobehavioral functions, neuroimaging, and quality of life for newly-diagnosed patients with primary CNS lymphoma at our institute. According to our cancer center, it is estimated that there would be around 25 cases of newly-diagnosed primary CNS lymphoma at our institute every year. By virtue of multidisciplinary management and teamwork consisting of neurosurgery, hematology, radiation oncology, neuroimaging expertise, and surgical pathology, investigators will attempt to recruit all potentially eligible patients with newly-diagnosed primary CNS lymphoma. Most importantly, the neuropsychologists will participate in our research project, in an effort to integrate the neurobehavioral outcomes into this prospective study. Accordingly, a battery of neuropsychological measures is used to evaluate neurobehavioral functions for the studied patients. The battery is composed of ten standardized neuropsychological tests, covering four domains sensitive to disease and treatment effects (executive function, attention, verbal memory, psychomotor speed), and QoL questionnaires.

Expected results. This prospective cohort study aims to explore and evaluate patients with PCNSL who are newly-diagnosed by using a standard battery of neurobehavioral functions plus neuroimaging studies. It is anticipated investigators will investigate and correlate neurotoxicity indicators in newly-diagnosed patients with PCNSL who are treated with cranial radiotherapy combined with or without MTX-based chemotherapy according to the multidisciplinary treatment guidelines implemented at a single institute.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histopathologic diagnosis of non-Hodgkin's lymphoma (NHL) by brain biopsy
* A typical MRI/CT scan for primary CNS lymphoma is defined as the presence of hypo, iso, or hyperintense parenchymal contrast-enhancing (usually homogeneously) mass lesion(s)
* Patients must have a normal or negative pre-treatment systemic evaluation including: i. A bone marrow aspirate and biopsy ii. CT scans of the chest, abdomen and pelvis iii. Patients must have adequate bone marrow reserve
* Patients must be HIV-1 negative
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for six months after completion of treatment

Exclusion Criteria:

* A past history of major psychiatric disease
* Prior cranial irradiation for any reasons
* Other active primary cancer with the exception of basal cell carcinoma of skin and cervical carcinoma in situ
* Pre-existing immunodeficiency such as renal transplant recipient

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly-diagnosed patients with primary CNS lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in neurocognitive functions from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Trail Making Test.
The change in memory functions from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Word Sequence Learning Test.
The change in general cognitive functions from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Mini Mental Status Examination.
The change in attention functions from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Paced Auditory Serial Addition Test-Revised
The change in executive functions from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Modified Card Sorting Test.
The change in verbal fluency from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Semantic association of verbal fluency.
The change in Intelligence from baseline up to 4 months after completing all courses of chemoradiation. | one week before the WBRT course, up to 4 months after completing all courses of chemoradiation
  Neurocognitive assessment including :
  Wechsler Adult Intelligence Scale (WAIS-III-R).

SECONDARY OUTCOMES:
The time from the date of recruitment to that of intracranial progression/failure noted on brain MRI | Baseline before the WBRT course; 2 months after completing all courses of chemoradiation, and then 4 months later.
Depression Inventory questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and then 4 months later.
  Questionnaires include:
  Beck Depression Inventory.
Anxiety Inventory questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and then 4 months later.
  Questionnaires include:
  Beck Anxiety Inventory.
Self- Evaluation questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and then 4 months later.
  Questionnaires include:
  National Taiwan University Irritability Scale Self- Evaluation (NTUIS-Self).
Family Evaluation questionnaires. | Baseline before the WBRT course; one month after completing the WBRT course; 2 months after completing all courses of chemoradiation, and then 4 months later.
  Questionnaires include:
  National Taiwan University Irritability Scale-Family Evaluation (NTUIS-Family).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan